# Manual of Procedures/Protocol

**Title**: A Double-Blind Randomized Placebo-Controlled Clinical Trial of Preoperative Gabapentin Prior to Vaginal Apical Suspension Prolapse Procedures

Fellow: Colin Johnson, MD PGY5

Research Mentor: Joseph Kowalski, MD

University of Iowa Hospitals and Clinics Department of Female Pelvic Medicine and Reconstructive Surgery Iowa City, IA July 2022 (Title page added June 25<sup>th</sup>, 2025)

#### INFORMED CONSENT DOCUMENT

Project Title: A Double-Blind Randomized Placebo-Controlled Clinical Trial of Preoperative Gabapentin Prior to Vaginal Apical Suspension Prolapse Procedures

**Principal Investigator:** Joseph Kowalski

**Research Team Contact:** Colin Johnson, colin-johnson@uiowa.edu, 319-384-8218

This consent form describes the research study to help you decide if you want to participate. This form provides important information about what you will be asked to do during the study, about the risks and benefits of the study, and about your rights as a research subject.

- If you have any questions about or do not understand something in this form, you should ask the research team for more information.
- You should discuss your participation with anyone you choose such as family or friends.
- Do not agree to participate in this study unless the research team has answered your questions and you decide that you want to be part of this study.

## WHAT IS THE PURPOSE OF THIS STUDY?

This is a research study. We are inviting you to participate in this research study because you are scheduled to have a vaginal procedure for uterine or vaginal prolapse.

The purpose of this research study is to determine if a one-time dose of the medication gabapentin just before surgery will help with pain after surgery. Notably this medication is commonly used for this but the data is mixed on whether it is effective.

Gabapentin is considered investigational, which means that it has not been approved by the U.S. Food and Drug Administration as it will be used in this study." Gabapentin is only FDA approved for seizures and postherpetic neuralgia (pain after a Shingles infection). Gabapentin is being compared to placebo in this study.

### **HOW MANY PEOPLE WILL PARTICIPATE?**

Approximately 110 people will take part in this study conducted by investigators at the University of Iowa.

### **HOW LONG WILL I BE IN THIS STUDY?**

If you agree to take part in this study, your involvement will last for roughly 48 hours (starting from administration of the medication just prior to the surgery until 24 hours after the surgery).

### WHAT WILL HAPPEN DURING THIS STUDY?

If you agree to take part in this study, you will receive the study medication in the preoperative area prior to your surgery. You will be randomly assigned to receive either a placebo (microcrystalline

cellulose) or gabapentin 300 mg. This means that whichever study treatment you receive will be determined purely by chance, like flipping a coin. Neither you nor the research team will know which study treatment you are receiving, but we will be able to get this information quickly if we need it to ensure your safety.

You will also receive acetaminophen and celecoxib (a medication similar to ibuprofen) per standard protocol. You will then undergo your planned procedure as normal. Your postoperative pain will be recorded in the postoperative area per usual hospital protocol. Between 24 and 36 hours after the surgery you will be verbally asked (in the hospital or over the phone if you have been discharged) a few questions regarding your pain control and other symptoms since surgery. This will take less than 5 minutes.

We will collect information about you from the electronic medical record including but not limited to demographics, medical histories, and postoperative pain scores. This information will be stored in a secure database and only identifiable with your unique study ID number.

## **Data Storage for Future Use**

Your information/data collected as part of this research study, even if identifiers are removed, will not be used or distributed for future research studies.

#### WHAT ARE THE RISKS OF THIS STUDY?

You may experience one or more of the risks indicated below from being in this study. In addition to these, there may be other unknown risks, or risks that we did not anticipate, associated with being in this study.

One risk of this study includes loss of confidentiality of protected health information (PHI).

You may receive a placebo (an inactive substance) during this study. This means that you would receive no active study treatment while participating and your postoperative pain could potentially be worse.

Other risks of this study include the risks of taking a one-time dose of 300 mg gabapentin. Notably in 2019, the U.S. Food and Drug Administration issued a warning that serious breathing difficulties may occur in patients using gabapentin or pregabalin in patients with respiratory risk factors and is now requiring that warnings about the risk of respiratory depression be added to the prescribing information of gabapentinoids. Respiratory depression has not been reported with a one-time low dose (300 mg) of gabapentin. See other risks below:

# <u>Likely / Common (more than 35%)</u>

Life Threatening: None

Serious: none Mild: none

### Less Likely / Less Common (10% - 35%)

Life Threatening: None

Serious: None

Mild: Dizziness, somnolence, gait disturbance

#### Rare (less than 10%)

Life Threatening: None

Serious: Respiratory depression

Mild: Visual disturbance, allergic reaction, nausea, vomiting

## WHAT ARE THE BENEFITS OF THIS STUDY?

You will not benefit directly from being in this study. However, we hope that, in the future, other people might benefit from this study because we will learn whether or not gabapentin is efficacious at decrease post-operative pain.

## WILL IT COST ME ANYTHING TO BE IN THIS STUDY?

You will not have any costs for being in this research study.

### WILL I BE PAID FOR PARTICIPATING?

You will not be paid for being in this research study.

## WHO IS FUNDING THIS STUDY?

The University and the research team are receiving no payments from other agencies, organizations, or companies to conduct this research study.

### WHAT IF I AM INJURED AS A RESULT OF THIS STUDY?

- If you are injured or become ill from taking part in this study, medical treatment is available at the University of Iowa Hospitals and Clinics.
- The University of Iowa does not plan to provide free medical care or payment for treatment of any illness or injury resulting from this study unless it is the direct result of proven negligence by a University employee.
- If you experience a research-related illness or injury, you and/or your medical or hospital insurance carrier will be responsible for the cost of treatment.

## WHAT ABOUT CONFIDENTIALITY?

We will keep your participation in this research study confidential to the extent permitted by law. However, it is possible that other people such as those indicated below may become aware of your participation in this study and may inspect and copy records pertaining to this research. Some of these records could contain information that personally identifies you.

- federal government regulatory agencies,
- the U.S. Food and Drug Administration
- auditing departments of the University of Iowa, and
- NuCara Pharmacy

• the University of Iowa Institutional Review Board (a committee that reviews and approves research studies)

To help protect your confidentiality, we will maintain records on a secure password protected local server (REDCAP) in-order-to minimize this risk. In addition, data forms will not contain any patient names or other personal information. Each form will contain only a unique subject identifier. Any paper data (deidentified) will be kept in a locked file cabinet in a locked office. If we write a report or article about this study or share the study data set with others, we will do so in such a way that you cannot be directly identified.

The University of Iowa Hospitals and Clinics generally requires that we document your participation in research occurring in a University of Iowa Health Care facility. This documentation will be in either your medical record or a database maintained on behalf of the institution reflecting that you are participating in this study. The information included will provide contact information for the research team as well as information about the risks associated with this study. We will keep this Informed Consent Document in our research files; it will not be placed in your medical record chart.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. A copy of the informed consent document will be available on this website. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

## WILL MY HEALTH INFORMATION BE USED DURING THIS STUDY?

The Federal Health Insurance Portability and Accountability Act (HIPAA) requires the University of Iowa Health to obtain your permission for the research team to access or create "protected health information" about you for purposes of this research study. Protected health information is information that personally identifies you and relates to your past, present, or future physical or mental health condition or care. We will access or create health information about you, as described in this document, for purposes of this research study. Once the University of Iowa Health has disclosed your protected health information to us, it may no longer be protected by the Federal HIPAA privacy regulations, but we will continue to protect your confidentiality as described under "Confidentiality."

We may share your health information related to this study with other parties including federal government regulatory agencies, the University of Iowa Institutional Review Boards and support staff, NuCara Pharmacy, and the University of Iowa Investigational Pharmacy.

You cannot participate in this study unless you permit us to use your protected health information. If you choose *not* to allow us to use your protected health information, we will discuss any non-research alternatives available to you. Your decision will not affect your right to medical care that is not research related. Your signature on this Consent Document authorizes the University of Iowa Health to give us permission to use or create health information about you.

Although you may not be allowed to see study information until after this study is over, you may be given access to your health care records by contacting your health care provider. Your permission for us

to access or create protected health information about you for purposes of this study has no expiration date. You may withdraw your permission for us to use your health information for this research study by sending a written notice to Joseph Kowalski (200 Hawkins Dr. Iowa City IA 52245, joseph-kowalski@uiowa.edu, 319-384-8218). However, we may still use your health information that was collected before withdrawing your permission. Also, if we have sent your health information to a third party, such as the study sponsor, or we have removed your identifying information, it may not be possible to prevent its future use. You will receive a copy of this signed document.

## **IS BEING IN THIS STUDY VOLUNTARY?**

Taking part in this research study is completely voluntary. You may choose not to take part at all. If you decide to be in this study, you may stop participating at any time. If you decide not to be in this study, or if you stop participating at any time, you won't be penalized or lose any benefits for which you otherwise qualify.

## Will I Receive New Information About the Study while Participating?

If we obtain any new information during this study that might affect your willingness to continue participating in the study, we'll promptly provide you with that information.

# Can Someone Else End my Participation in this Study?

Under certain circumstances, the researchers might decide to end your participation in this research study earlier than planned. This might happen because in our judgement it would not be safe for you to continue.

## WHAT IF I HAVE QUESTIONS?

We encourage you to ask questions. If you have any questions about the research study itself, please contact: Joseph Kowalski or Colin Johnson (319-384-8218). If you experience a research-related injury, please contact Joseph Kowalski or Colin Johnson (319-384-8218).

If you have questions, concerns, or complaints about your rights as a research subject or about research related injury, please contact the Human Subjects Office, 105 Hardin Library for the Health Sciences, 600 Newton Rd, The University of Iowa, Iowa City, IA 52242-1098, (319) 335-6564, or e-mail <a href="mailto:irb@uiowa.edu">irb@uiowa.edu</a>. General information about being a research subject can be found by clicking "Info for Public" on the Human Subjects Office web site, <a href="http://hso.research.uiowa.edu/">http://hso.research.uiowa.edu/</a>. To offer input about your experiences as a research subject or to speak to someone other than the research staff, call the Human Subjects Office at the number above.

This Informed Consent Document is not a contract. It is a written explanation of what will happen during the study if you decide to participate. You are not waiving any legal rights by signing this Informed Consent Document. Your signature indicates that this research study has been explained to you, that your questions have been answered, and that you agree to take part in this study. You will receive a copy of this form.

| Subject's Name (printed): | |
|---|---|
| (Signature of Subject) | (Date) |
| Statement of Person Who Obtained Cons | <u>ent</u> |
| - | ubject or, where appropriate, with the subject's legally that the subject understands the risks, benefits, and is research study. |
| (Signature of Person who Obtained Consent | (Date) |